CLINICAL TRIAL: NCT03507140
Title: Biliary and Intestinal Microbiota Study in Liver Transplanted Patients
Brief Title: Microbiota Study in Liver Transplanted Patients
Acronym: BIM-LT
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.332
Record Dates: First submitted 2018-04-05; First posted 2018-04-24 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma; Liver Transplant; Microbiota
Keywords: cirrhosis; hepatocellular carcinoma; Liver transplantation; Microbiota
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bile, blood, saliva, feces and urine in donor and recipients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multiple sampling — Bile, saliva, feces, urine et blood samples before and after liver transplantation in recipients.
  Bile, saliva, feces, urine et blood samples during liver removal in donors.

SUMMARY:
Many studies describe the relationship between microbiota alteration and the occurrence of metabolic, alcoholic or inflammatory liver diseases. Nevertheless, the modifications of microbiota during liver transplantation (LT) as well as its implication are poorly studied. Similarly, only the intestinal microbiota is studied in this context, and no data are available on the biliary microbiota, even if it is known that bile microbiota can interfere with hepatobiliary diseases.

This study proposes a clinical and biological in-depth follow-up with multiple sampling of liver transplanted patients to study biliary and intestinal microbiota alterations along LT, as well as bile acids metabolism in corresponding fluids.

Indeed, in recipient samples as saliva, blood, urine, and feces can be taken before LT, and surgeons can easily perform bile sampling during LT. In donors all samples can be taken during liver removal. This offers the opportunity to have a microbiotic landscape of individuals without liver disease (donor), and patients suffering from a chronic liver disease or a liver cancer before and after transplantation.

Also, in Grenoble University hospital, in case of biliary anastomotic incongruence, a biliary stent is placed during LT in 60% of recipients. This stent is removed by endoscopic retrograde cholangiopancreatography (ERCP) within 6 months after LT, offering a second opportunity to obtain bile samples in transplanted patients, after the early post-LT period. Patients who do not require a biliary stent will also be included for the study of secondary objectives, as intestinal microbiota is very poorly characterized in liver transplanted patients too. A portion of the patients without biliary stent, may also develop an anastomotic biliary stricture requiring an ERCP. If this ERCP is realized within the follow-up period of the study, the patient will also be included in the primary objective of the study.

These multiple and sequential samples will allow a complete analysis of microbiota changes in LT patients and aim to answer to 3 questions:

1. What are the modifications of intestinal and biliary microbiomes during LT?
2. What is the influence of bile acids' composition on intestinal and biliary microbiota?
3. What are the relationships between microbiome alterations and the emergence of LT complications?

ELIGIBILITY:
Inclusion Criteria:

Recipients:

* Age ≥ 18 years old
* Absence of LT contraindications
* Patient undergoing liver transplantation
* Patient legally able to give written consent.
* Person affiliated to social security

Donors:

Cadaveric-donor liver transplantation

Exclusion Criteria:

* Living-related liver transplantation
* LT contraindications
* All subjects protected by articles L1121-5 and L1121-8 of French public health law (Subject under administrative or judicial control, person who are protected under the act, person hospitalized without their consent, prisoners and pregnant or breast-feeding women).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered on the waiting list fo liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Comparison of the relative abundance of pathobionts and symbionts before and 6 months after liver transplantation, in the bile of recipients. | During LT and 6 months after LT
  Beneficial bacterias/pathobionts ratio before and 6 months after liver transplantation in the bile of recipients.

SECONDARY OUTCOMES:
Comparison of the relative abundance of pathobionts and beneficial bacteria at the time, and 6 months after liver transplantation, in the feces of recipients. | Before LT (6 months maximum) and 6 months after LT
  Intestinal beneficial bacterias/pathobionts ratio before and 6 months after liver transplantation in recipients.
Comparison of bile microbial diversity at the time, and 6 months after liver transplantation, in LT recipients. | During LT and 6 months after LT
  Proportion of the different microbial populations in recipients' bile.
Comparison of fecal microbial diversity before, and 6 months after liver transplantation, in LT recipients. | Before LT (6 months maximum) and 6 months after LT
  Proportion of the different microbial populations in recipients' feces.
Study the correlation between bile microbiota of donors and recipients after LT. | During LT and 6 months after LT
  Proportion of the different biliary microbial populations of donors and in their corresponding recipient.
Study the correlation between fecal microbiota of donors and recipients after LT. | Before LT (6 months maximum) and 6 months after LT
  Proportion of the different intestinal microbial populations of donors and their corresponding recipient.
Study the relationships between bile microbiota changes and intestinal microbiota modifications in recipients, before and after LT. | Before LT (6 months maximum) and 6 months after LT
  Correlation between microbial populations' proportions in bile and in feces in donors and in recipients.
Study the modifications of bile acid profiles in recipients between before and after LT. | Before LT (6 months maximum) and 6 months after LT
  Proportions of total, primary and secondary biles acids in urine, feces and bile of donors and recipients.
Study the influence of bile acids'composition on bile microbiota along transplantation. | Before LT (6 months maximum) and 6 months after LT
  Correlation between the evolution of pathobionts and beneficial bacterias' proportions in bile and the different bile acids (BA) profiles (proportions of primary and secondary BAs).
Study the influence of bile acids' composition on intestinal microbiota along transplantation. | Before LT (6 months maximum) and 6 months after LT
  Correlation between the evolution of pathobionts and beneficial bacterias' proportions in feces and the different bile acids profiles (proportions of primary and secondary BAs) before and after LT.
Study the relationships between microbiota and the emergence of LT complications (post LT infections, acute liver allograft reject, etc). | Before LT (6 months maximum) and 6 months after LT
  Correlation between the evolution of pathobionts and beneficial bacterias' proportions in feces and the different bile acids profiles (proportions of primary and secondary BAs).
Biobanking of blood, saliva, bile, feces and urine for further analyses such as metabolomic studies on blood, urine and feces metagenomic studies on saliva, and immunomonitoring on blood. | Before LT (6 months maximum) and 6 months after LT

CONTACTS AND LOCATIONS:
Overall Officials: Gael ROTH, MD, Principal Investigator — GRENOBLE ALPES UNIVERSITY HOSPITAL
Locations (1):
- CHU de GRENOBLE ALPES, Grenoble, France

IPD SHARING:
Plan to Share IPD: No